CLINICAL TRIAL: NCT03988257
Title: The Effectiveness of Pleuran in Treatment of Acute Gastroenteritis in Children- a Randomized, Placebo-controlled, Double-blind Trial
Brief Title: The Effectiveness of Pleuran in Treatment of Acute Gastroenteritis in Children
Acronym: EPTAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Nutricia Foundation (Other); Pleuran, s.r.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5FNUT11; KB/45/2018 (Other: The Medical University of Warsaw Bioethical Committee)
Record Dates: First submitted 2019-06-14; First posted 2019-06-17 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2021-10

CONDITIONS: Diarrhoea;Acute
Keywords: Acute diarrhoea; Infectious diarrhoea; Pleuran; Beta-glucan; Duration of diarrhoea; Severity of diarrhoea; Randomized Controlled Trails as Topic
MeSH Terms: conditions — Dysentery

STUDY DESIGN:
Intervention Model Description: This will be a randomized, double-blind, placebo-controlled trial, with allocation 1:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients, their caregivers, researchers, physicians, nurses, the statistician will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Imunoglukan PH4 syrup (10 mg of pleuran and 10 mg of vitamin C in 1 ml of syrup) in a dose 1 ml / 5 kg body weight, once a day.
  Interventions: Dietary Supplement: Imunoglukan PH4
- Control group (Placebo Comparator): A vitamin C syrup (10 mg of vitamin C in 1 ml of syrup) in a dose 1 ml / 5 kg body weight.
  Interventions: Dietary Supplement: Placebo (vitamin C syrup)

INTERVENTIONS:
Dietary Supplement: Imunoglukan PH4 — Children allocated to experimental group will receive Imunoglukan PH4 syrup (10 mg of pleuran and 10 mg of vitamin C in 1 ml of syrup) in a dose 1 ml / 5 kg body weight, once a day in the morning, before the first meal, until signs of AGE subside (< 3 stools / 24 hours and normalization of stool consistency - grade 2-5 according to Bristol Stool Form Scale) or until the 14th day of the intervention.
  Arms: Experimental group
Dietary Supplement: Placebo (vitamin C syrup) — Children allocated to control group will receive a placebo: a vitamin C syrup (10 mg of vitamin C in 1 ml of syrup) in a dose 1 ml / 5 kg body weight, once a day in the morning, before the first meal, until signs of AGE subside (< 3 stools / 24 hours and normalization of stool consistency - grade 2-5 according to Bristol Stool Form Scale) or until the 14th day of the intervention.
  Arms: Control group

SUMMARY:
Acute gastroenteritis (AGE) is one of the most common causes of children's morbidity and mortality globally. Oral or intravenous rehydration is the only effective treatment in reducing morbidity and mortality rates in AGE. However, new attempts to identify other therapeutic methods to reduce the symptoms of diarrhea are of interest. The administration of pleuran (β- (1,3 / 1,6) -D-glucan) appears to be such an alternative. In Poland, pleuran is being marketed for treating AGE. Its potential immunomodulatory effect is based on the stimulation of both humoral and cellular immunity. The active substance of the product (pleuran) was extracted by unique and patented technology from Pleurotus ostreatus. The substance was previously isolated, identified and chemically characterized by Karacsonyi and Kunia. Pleuran is registered as a diet supplement and distributed in 20 European and non-European countries. The testing for toxicity was performed by the Institute of Preventive and Clinical Medicine of Slovak Medical University (Final Report No. 5-51/04) and the tests were performed in compliance with the criteria of the Directive of Good Laboratory Practice and Directive 2004/10/EC of the European Parliament and the Council of 11th February 2004.

To evaluate the efficacy of pleuran in reducing the duration and the severity of AGE symptoms in children, a randomized, placebo-controlled, fully-blind study has been designed. A total of 120 children will be randomly assigned to receive either Imunoglukan PH4 syrup in the experimental group or matching placebo in the control group. The primary outcome measure will be the duration of diarrhea. The statistical analysis of the results will be conducted in both intention-to-treat and per-protocol approach.

DETAILED DESCRIPTION:
Study design: This will be a randomized, fully-blind, placebo-controlled trial, with allocation 1:1.

Study population: Children aged 13- 120 months, hospitalized or requiring a visit to the emergency department due to acute gastroenteritis (AGE) lasting at least 24 h, but no longer than 72 h at the time of inclusion to the study.

The setting of the study: The study participants will be recruited from patients requiring hospitalization in 4 paediatric departments or counselling in the emergency department (ED) due to AGE in the Paediatric Teaching Clinical Hospital, the Medical University of Warsaw.

Pre-intervention assessment:

We will evaluate the inclusion and exclusion criteria of the study within 24 hours of hospitalization or ED visit basing on the physical examination and interviews with caregivers. The BMI will be calculated and put on WHO percentiles charts. In order to determine the etiology of AGE, the stool sample will be collected for viral tests (rota-, adeno- and noroviruses markers) before the intervention. If any indication for microbiological stool investigation occurs (the patient in severe condition or with prolonged symptoms in whom specific treatment is considered, or patient with underlying chronic disease), the stool sample will be cultured. The caregivers will be informed about the purpose, methods, safety of the intervention and the course of the study. In order to ensure that the assessed parameters and endpoints are comparable appropriate scales will be applied. To assess the severity of diarrhea, the Modified Vesikari Score will be used. The dehydration degree will be evaluated by means of the WHO scale and the Clinical Dehydration Scale (CDS) recommended by the European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN). The Bristol Stool Form Scale will help to objectify the assessment of stool consistency.

Randomization:

The randomization will involve the random allocation of patients to group A or B. The stratified randomization has been designed with the use of two subgroups. The subgroups will be created depending on the duration of diarrhea at the time of enrolment: 24-48 h (short-lasting diarrhea- SLD) and 48-72 h (long-lasting diarrhea- LLD). The participants of each subgroup will be randomly allocated to the study groups (experimental or control), in blocks of four.

Allocation concealment and blinding:

The active product and placebo will be prepared, weighed, packaged in identical bottles and signed with random numbers by the manufacturer, with the blinded meaning of numbers. The information about the allocation will be deposited in a sealed envelope in a safe place in the administrative part of the department, kept by the independent person not involved in the study. The study product will be delivered to the main researcher in boxes of four, ensuring the contest of 2 active and 2 placebo samples in each box. Subsequent boxes will be used to allocate consecutive patients within the subgroups A and B. By opening each subsequent box, the numbers of bottles in the box will be randomly assigned to the next four patients in a subgroup by the researcher. The contents of the bottles will look and taste the same. Researchers, caregivers, patients, and a person responsible for the statistical analysis will be blinded to the intervention until the completion of the study.

Intervention:

Children allocated to the experimental group will receive Imunoglukan PH4 oral suspension (10 mg of pleuran and 10 mg of vitamin C in 1 ml of syrup) in a dose 1 ml / 5 kg body weight, while patients in the control group will receive a placebo: a vitamin C oral suspension (10 mg of vitamin C in 1 ml of syrup) in a dose 1 ml / 5 kg body weight. Both syrups will be administered once a day in the morning, before the first meal, until signs of AGE subside (< 3 stools / 24 hours and normalization of stool consistency - grade 2-5 according to Bristol Stool Form Scale) or until the 14th day of the intervention.

Concomitant treatment:

To ensure proper rehydration, patients in both groups will receive an oral rehydration solution (ORS) or intravenous fluids if necessary, according to daily fluids requirements. A normal diet will be delivered. Each patient will receive antipyretic, analgesic (Ibuprofen, Acetaminophen), and antiemetic (Ondansetron) if necessary. Patients will not receive other medicines that may interfere with the disease course (probiotics, Diosmectite, Racecadotril). If indications occur, the patient will receive an antibiotic according to the ESPGHAN recommendations

Follow up:

During hospitalization, patients will be examined every day by the physician, with the assessment of dehydration level, the need for intravenous rehydration or concomitant treatment. The results of the evaluation will be recorded in the Case Report Form (CRF). Both during and after the hospitalization, the caregiver will record AGE symptoms in a diary (a number of stools per day, their consistency and accompanying symptoms e.g. fever, vomiting, abdominal pain). Complete diaries will be collected from caregivers via email or by telephone conversation. After discharge, caregivers will have the possibility to contact a physician to receive basic consultation about oral rehydration and eventual side effects.

Data management:

Coded, paper CRF containing all the scales and questionnaires will be created for each patient. After finishing the observation, the data from the symptoms diaries completed by the caregivers will be transferred by the physician to the paper versions of the CRFs. After completing the study, data from the CRFs will be transferred to two electronic databases by two independent persons to confirm the accuracy of the data. Electronic database and CRFs will be prepared in Statistical Analysis System (SAS) software. The collected data will be properly stored to allow for data verification. Confidentiality of data, including personal data of the study participants, will be maintained.

Adverse events (AE) Every AE will be recorded and reported to the investigator and manufacturer, according to a pre-established procedure.

Sample size:

The Altman nomogram was used to estimate the sample size of experimental and control groups. To demonstrate a clinically relevant difference of 24 h in duration of AGE symptoms in experimental and control groups, with 5% significance level and a power of 90%, assuming the standard deviation of the variable in each group of 40 h, a sample of 110 patients will be needed (55 patients in each group). Allowing for 10% attrition of participants during the study, we estimated the sample size as 120 patients (60 patients for each experimental and control group).

Statistical analysis:

Descriptive statistics will be used to summarise baseline characteristics. Intention-to-treat (ITT) and per protocol analyses will be used to present the results of the study. The comparison of group A and B in terms of the primary endpoint (duration of diarrhea) will be performed with Student's t-test if the p-value of the Shapiro-Wilk test will be >0.05. Otherwise, the Mann-Whitney U test will be used. In the case of dropouts or not completed observations before the 14th days of the study, the log-rank test will be performed. The Chi-squared test or Fisher's exact test will be used to compare the groups A and B in terms of the incidence of adverse events and the severity of diarrhea. Statistical significance will be based on two-tailed tests with p-value of 5%. All estimates will be presented with 95% confidence interval.

Amendment No 1:

The presented protocol contains amendments approved by the Bioethics Committee on May 11, 2020. The main reason for those changes was an unsatisfactory pace of recruitment in the first 11 months of study commencement. A detailed analysis revealed the reduction in the number of hospitalizations due to AGE in our Department compared to the previous year and difficulties in meeting the inclusion criteria. In the following months, the COVID pandemic significantly limited the number of patients hospitalized in our hospital. By the time the changes were made we recruited only three patients into the study.

For the listed reasons we have introduced the following changes to the protocol:

1. The first version of the protocol assumed the recruitment of patients among hospitalized children only. The amendment introduced the possibility of recruitment also among children requiring counselling in the emergency department.
2. Initially, patients were recruited only at the Department of Pediatric with Clinical Assessment Unit (the unit initiating and conducting the study). The amendment introduced 4 other clinics of the Pediatric Teaching Clinical Hospital, the Medical University of Warsaw, including the Emergency Department.
3. The age group of recruited patients initially 13- 60 months (up to 6 years of age) was extended to older children 13- 120 months (up to 10 years of age).

Amendment No 2

The presented protocol contains amendments approved by the Bioethics Committee on December 13, 2021. The main reason for those changes was an unsatisfactory pace of recruitment, caused by a significant change in the profile of hospitalized patients due to the SARS-CoV2 pandemic. By the time the changes were made we recruited only ten patients into the study.

1. The amendment introduced two other locations for patient recruitment: The Department of Pediatrics of Warsaw Children's Hospital and The Department of Pediatrics of Hospital of Trzebnica, Poland.
2. The amendment introduced the possibility of recruitment among children requiring outpatient counseling due to acute diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 13-120 months, hospitalized or requiring a visit in the emergency department (ED) or outpatient consultation due to AGE, defined as a decrease in the stool consistency (grade 6 or 7 in Bristol Stool Form Scale) and/or an increase in the frequency of stool evacuations > 3 in 24 hours.
* Duration of symptoms 24-72 hours at the time of inclusion.
* Caretaker's written, informed consent.

Exclusion Criteria:

* Duration of symptoms > 72 hours at the time of inclusion.
* Co-occurring other systemic infectious diseases (ex. pneumonia, sepsis).
* Diagnosed immune deficiency.
* Malnutrition (defined as the body mass index (BMI) <-2 SDS (Standard Deviation Scores) or < 3rd percentile based on the World Health Organization (WHO) percentile charts.
* Chronic diarrhoeal gastrointestinal disease (inflammatory bowel disease, short bowel syndrome, cystic fibrosis, celiac disease, food allergy).
* Use of antibiotics, probiotics, prebiotics or anti-diarrhea (Diosmectite, Racecadotril) medicines within 7 days prior to enrolment into the study.
* Use of probiotics, Diosmectite, Racecadotril during the current AGE episode.
* Use of pleuran in the 14 days prior to enrolment into the study.
* Parallel involvement of the patient in other clinical trials, with the exception of observational studies.
* No legal caregivers' consent to participate in the study

Ages: 13 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The duration of diarrhoea. | Daily assessment, by the physician and/ or the patient's caregiver during until the 14th day of observation
  The duration of diarrhoea, defined as the time (hours) until normalization of stool consistency (grade 2, 3, 4 or 5 according to Bristol Stool Form Scale) and until normalization of number of stools per day.

SECONDARY OUTCOMES:
The duration of hospitalization. | Daily assessment until the 14th day of observation.
  The length of hospital stay due to AGE (number of days).
The number of days with need for intravenous rehydration. | Daily assessment until the discharge from hospital.
  The need for intravenous rehydration will be assessed daily by physician, based on CDC (Centers for Disease Control and Prevention) and WHO dehydration scales.
The number of hours until normalization of stools consistency ( type 2-5 according to Bristol Stool Consistency Scale). | Daily assessment until the 14th day of observation.
  Assessed on the basis of the diary completed by the physician and the caregiver.
The number of hours until the normalization of number of stools per day (<3 stools/ day). | Daily assessment until the 14th day of observation.
  Assessed on the basis of the diary completed by the physician and the caregiver.
The percentage of children with moderate and severe diarrhea. | Assessed after the 14th day of the observation.
  Assessed by the Modified Vesikari Scale in the end of observation.
The time until the improvement of the child's general condition according to the caregiver's assessment. | Daily assessment until the 14th day of observation.
  Based on the caregiver assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Kuchar, MD PhD, Study Chair — The Department of Pediatrics with Clinical Assessment Unit, The Medical University of Warsaw
Locations (1):
- The Department of Pediatrics with Clinical Assessment Unit, The Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
The Study protocol will be publicly available during the Study commencement. Other documents (Statistical Analysis Plan, Clinical Research Form, Informed Consent Form) will be available on request from authorized institutions.
  Individual deidentified participant data will be available upon reasonable request for researchers who provide a methodologically sound proposal that has been approved by an independent bioethical committee. This will be available immediately after study result publication, for a minimum of 5 years. To gain access, data requestors will need to sign a data access agreement.
  Additionally, The Medical University of Warsaw committed to share with PLEURAN s.r.o. an unprocessed, deidentified participant data obtained during the Study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Documents listed above will be available during the Study commencement, while individual deidentified participant data after the Study results publication, for a minimum of 5 years.
Access Criteria: The study protocol will be publicly available. Other documents listed above (Statistical Analysis Plan, Clinical Research Form, Informed Consent Form) will be available on request for medical journal editors, The Bioethical Committee of The Medical University of Warsaw, and the Study Primary Sponsor (The Medical University of Warsaw) for the purpose of the Study methodology and ethics monitoring.

REFERENCES:
- [Background] Guarino A, Ashkenazi S, Gendrel D, Lo Vecchio A, Shamir R, Szajewska H; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition; European Society for Pediatric Infectious Diseases. European Society for Pediatric Gastroenterology, Hepatology, and Nutrition/European Society for Pediatric Infectious Diseases evidence-based guidelines for the management of acute gastroenteritis in children in Europe: update 2014. J Pediatr Gastroenterol Nutr. 2014 Jul;59(1):132-52. doi: 10.1097/MPG.0000000000000375. PMID 24739189
- [Background] Freedman SB, Ali S, Oleszczuk M, Gouin S, Hartling L. Treatment of acute gastroenteritis in children: an overview of systematic reviews of interventions commonly used in developed countries. Evid Based Child Health. 2013 Jul;8(4):1123-37. doi: 10.1002/ebch.1932. PMID 23877938
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Diarrhoea and Vomiting Caused by Gastroenteritis: Diagnosis, Assessment and Management in Children Younger than 5 Years. London: RCOG Press; 2009 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK63844/ PMID 22132432
- [Background] Hojsak I, Fabiano V, Pop TL, Goulet O, Zuccotti GV, Cokugras FC, Pettoello-Mantovani M, Kolacek S. Guidance on the use of probiotics in clinical practice in children with selected clinical conditions and in specific vulnerable groups. Acta Paediatr. 2018 Jun;107(6):927-937. doi: 10.1111/apa.14270. Epub 2018 Apr 16. PMID 29446865
- [Background] Szajewska H, Guarino A, Hojsak I, Indrio F, Kolacek S, Shamir R, Vandenplas Y, Weizman Z; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition. Use of probiotics for management of acute gastroenteritis: a position paper by the ESPGHAN Working Group for Probiotics and Prebiotics. J Pediatr Gastroenterol Nutr. 2014 Apr;58(4):531-9. doi: 10.1097/MPG.0000000000000320. PMID 24614141
- [Background] van den Berg J, Berger MY. Guidelines on acute gastroenteritis in children: a critical appraisal of their quality and applicability in primary care. BMC Fam Pract. 2011 Dec 2;12:134. doi: 10.1186/1471-2296-12-134. PMID 22136388
- [Background] Di Luzio NR. Update on the immunomodulating activities of glucans. Springer Semin Immunopathol. 1985;8(4):387-400. doi: 10.1007/BF01857392. No abstract available. PMID 4089757
- [Background] Chan GC, Chan WK, Sze DM. The effects of beta-glucan on human immune and cancer cells. J Hematol Oncol. 2009 Jun 10;2:25. doi: 10.1186/1756-8722-2-25. PMID 19515245
- [Background] Jesenak M, Majtan J, Rennerova Z, Kyselovic J, Banovcin P, Hrubisko M. Immunomodulatory effect of pleuran (beta-glucan from Pleurotus ostreatus) in children with recurrent respiratory tract infections. Int Immunopharmacol. 2013 Feb;15(2):395-9. doi: 10.1016/j.intimp.2012.11.020. Epub 2012 Dec 20. PMID 23261366
- [Background] Jesenak M, Urbancek S, Majtan J, Banovcin P, Hercogova J. beta-Glucan-based cream (containing pleuran isolated from pleurotus ostreatus) in supportive treatment of mild-to-moderate atopic dermatitis. J Dermatolog Treat. 2016 Aug;27(4):351-4. doi: 10.3109/09546634.2015.1117565. Epub 2015 Dec 10. PMID 26654776
- [Background] Bobovcak M, Kuniakova R, Gabriz J, Majtan J. Effect of Pleuran (beta-glucan from Pleurotus ostreatus) supplementation on cellular immune response after intensive exercise in elite athletes. Appl Physiol Nutr Metab. 2010 Dec;35(6):755-62. doi: 10.1139/H10-070. PMID 21164546
- [Background] Bergendiova K, Tibenska E, Majtan J. Pleuran (beta-glucan from Pleurotus ostreatus) supplementation, cellular immune response and respiratory tract infections in athletes. Eur J Appl Physiol. 2011 Sep;111(9):2033-40. doi: 10.1007/s00421-011-1837-z. Epub 2011 Jan 20. PMID 21249381
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Derived] Wzorek-Lyczko K, Piwowarczyk A, Wozniak W, Kuchar E, Szymanski H. A randomised trial of pleuran in paediatric acute gastroenteritis. Sci Rep. 2025 May 15;15(1):16912. doi: 10.1038/s41598-025-94893-3. PMID 40374943
- [Derived] Wzorek-Lyczko K, Piwowarczyk A, Kuchar E. Protocol of the study: the effectiveness of pleuran in the treatment of acute gastroenteritis in children-a randomised, placebo-controlled, double-blind trial (EPTAGE). BMJ Open. 2021 Mar 11;11(3):e042370. doi: 10.1136/bmjopen-2020-042370. PMID 33707267